CLINICAL TRIAL: NCT00142558
Title: A Randomized, Double-Blind, Active-Comparator-Controlled 5-Day Trial of the Effect of Etoricoxib 120 mg Versus Indomethacin 150 mg in the Treatment of Acute Gout
Brief Title: A Study Evaluating the Effect of Etoricoxib and Indomethacin in the Treatment of Acute Gout (0663-081)(COMPLETED)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0663-081; MK0663-081; 2005_062
Record Dates: First submitted 2005-08-31; First posted 2005-09-02 (Estimated); Last update posted 2024-08-15 (Actual); Status verified 2022-02

CONDITIONS: Acute Gout
Keywords: Arcoxia
MeSH Terms: interventions — Etoricoxib; Duration of Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: MK0663; etoricoxib / Duration of Treatment: 5 Days
Drug: Comparator: indomethacin 75 mg sustained release capsule / Duration of Treatment: 5 Days

SUMMARY:
A study to evaluate the effects of etoricoxib and indomethacin in the treatment of acute gout.

ELIGIBILITY:
Inclusion Criteria:

* Males or females at least 18 years of age who have acute gout.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2005-01-01 (Actual); Primary Completion 2005-05-01 (Actual); Study Completion 2005-05-01 (Actual)

PRIMARY OUTCOMES:
Patient assessment of pain (0- to 4- Likert scale)

SECONDARY OUTCOMES:
Patient Global Assessment of Response to Therapy (0- to 4- point scale)
Investigator Global Assessment of Response to Therapy (0- to 4- point scale)
Tenderness of the study joint (0- to 3-point scale)
Swelling of the study joint (0- to 3-point scale)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Derived] Navarra S, Rubin BR, Yu Q, Smugar SS, Tershakovec AM. Association of baseline disease and patient characteristics with response to etoricoxib and indomethacin for acute gout. Curr Med Res Opin. 2007 Jul;23(7):1685-91. doi: 10.1185/030079907x210750. PMID 17588299